CLINICAL TRIAL: NCT01853982
Title: A Multicenter, Open-Label, Randomized Study to Compare the Safety and Efficacy of Intravenous Ceftolozane/Tazobactam With That of Piperacillin/Tazobactam in Ventilator Associated Pneumonia
Brief Title: Study of Intravenous Ceftolozane/Tazobactam Compared to Piperacillin/Tazobactam in Ventilator-Associated Pneumonia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated to focus on a larger study within the clinical development program.
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7625A-009; CXA-NP-11-08 (Other: Cubist Study Number)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Ventilator-Associated Pneumonia (VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — ceftolozane, tazobactam drug combination; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftolozane/Tazobactam (Experimental): 3000 milligrams (mg) ceftolozane/tazobactam (comprised of 2000 mg ceftolozane and 1000 mg tazobactam), administered intravenously (IV), every 8 hours for 8 days
  Interventions: Drug: Ceftolozane/Tazobactam
- Piperacillin/Tazobactam (Active Comparator): 4500 mg piperacillin/tazobactam (comprised of 4000 mg piperacillin and 500 mg tazobactam), administered IV, every 6 hours for 8 days
  Interventions: Drug: Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Ceftolozane/Tazobactam
  Arms: Ceftolozane/Tazobactam
Drug: Piperacillin/Tazobactam
  Other Names: Zosyn
  Arms: Piperacillin/Tazobactam

SUMMARY:
This is a Phase 3, multicenter, prospective, randomized, open-label, study to compare the safety and efficacy of intravenous (IV) ceftolozane/tazobactam with that of IV piperacillin/tazobactam in the treatment of ventilator-associated pneumonia (VAP) in adult participants .

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has received mechanical ventilation for > 48 hours
* Acute Physiology and Chronic Health Evaluation (APACHE) II score of 11-35
* Presence of a new or progressive infiltrate on chest x-ray
* Presence of clinical criteria consistent with VAP

Key Exclusion Criteria:

* History of moderate or severe hypersensitivity reactions to beta-lactam antibiotics
* Known end stage renal disease or requirement for dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-06-14 (Actual); Primary Completion 2013-11-20 (Actual); Study Completion 2013-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Obiamiwe Umeh, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (19):
- United States (11):
  - Jacksonville, Florida
  - Chicago, Illinois
  - Baltimore, Maryland
  - Duluth, Minnesota
  - Omaha, Nebraska
  - Jamaica, New York
  - The Bronx, New York
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Abington, Pennsylvania
  - Nashville, Tennessee
- Australia (5):
  - Herston, Queensland
  - Meadowbrook, Queensland
  - Nambour, Queensland
  - Southport, Queensland
  - Woolloongabba, Queensland
- New Zealand (3):
  - Auckland
  - Christchurch
  - Wellington

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On 31 Dec 2013, enrollment was closed and the CXA-NP-11-08 study was electively terminated by the Sponsor in order to devote all resources in initiating and completing the larger registrational study (CXA-NP-11-04), which was also being conducted as part of the clinical development program for nosocomial pneumonia.
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam | Piperacillin/Tazobactam
Started | 2 | 2
Received at Least 1 Dose of Study Drug | 2 | 2
Completed | 0 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ceftolozane/Tazobactam: 3000 mg ceftolozane/tazobactam (comprised of 2000 mg ceftolozane and 1000 mg tazobactam), administered IV, every 8 hours for 8 days
- Total: Total of all reporting groups
Arm/Group | Ceftolozane/Tazobactam | Piperacillin/Tazobactam | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0
  BTWN | 1 | 2 | 3
  GTE65 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at the End of Therapy Visit
Time Frame: 24 hours after last dose of study drug
Population: There is no analysis population or data available for this measure. This study was electively terminated to focus on a larger registrational study, which was also part of the clinical development program for nosocomial pneumonia.
Arm/Group | Ceftolozane/Tazobactam | Piperacillin/Tazobactam
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ceftolozane/Tazobactam | Piperacillin/Tazobactam
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam (N=2) | Piperacillin/Tazobactam (N=2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
CNS ventriculitis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane/Tazobactam (N=2) | Piperacillin/Tazobactam (N=2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was electively terminated to focus on a larger registrational study, which was also part of the clinical development program for nosocomial pneumonia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other